CLINICAL TRIAL: NCT03424421
Title: Anterior Shoulder Instability Treated with a Semitendinosus Subscapular Sling Procedure. Pilot Study, a New Surgical Procedure
Brief Title: Anterior Shoulder Instability Treated with a Semitendinosus Subscapular Sling Procedure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Møre og Romsdal HF (Other Government)
Collaborators: Norwegian University of Science and Technology (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/1292
Record Dates: First submitted 2018-01-26; First posted 2018-02-07 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Anterior Shoulder Dislocation; Joint Instability
Keywords: Shoulder Joint; Orthopedics; Arthroscopy
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Intervention Model Description: pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- subscapular sling (Experimental): semitendinosus subscapular sling procedure
  Interventions: Procedure: subscapular sling

INTERVENTIONS:
Procedure: subscapular sling — semitendinosus subscapular sling procedure

SUMMARY:
The arthroscopic subscapular sling procedure is a new technique for shoulder stabilization, which has been developed in human cadaveric studies by Klungsøyr et al, but has yet to be tested clinically. The procedure stabilizes the shoulder by using a semitendinosus graft that makes a new labrum and a sling around the subscapular tendon. Extensive biomechanical robotic testing of the procedure shows significant less translation and thus better stability of the humeral head with the sling compared to a normal Bankart repair. The investigators consider the biomechanical results after robotic testing sufficient to advocate a planned pilot study in humans. In this pilot study the clinical and radiological results of the sling will be investigated in a small number of cases. The safety of the subscapular sling procedure will be assessed. This studies results are expected to be a further step towards implementation of the sling procedure as a surgical option for shoulder instability.

ELIGIBILITY:
Inclusion Criteria:

* Clinical anterior instability of the shoulder and/or previous failed Bankart repair or arthroscopic findings concluding with too weak anterior structures to perform capsulolabral or labrum repair
* Be able to understand oral and written Norwegian /English

Exclusion Criteria:

* Cuff injury or previous cuff repair
* Surgical fracture treatment of the glenoid or humeral head
* Other instability procedures in the shoulder except Bankart repair and anterior capsular plications
* Previous infections in the shoulder
* MRI detectable fatty infiltration of the subscapularis or partial/total tendon rupture
* Severe glenohumeral arthrosis
* Multidirectional or posterior instability
* Not able to comply fully with the protocol due to psychosocial and physical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2032-08-30 (Estimated)

PRIMARY OUTCOMES:
The recurrence rate of shoulder dislocation after the subscapular sling | 2 , 5 and 10 years follow up.
  Explore to what extent the subscapular sling procedure is successful in preventing recurrent shoulder dislocations

SECONDARY OUTCOMES:
Changes in the Western Ontario Shoulder Instability index (WOSI) score | 2, 5 and 10 years follow up.
  Changes in the WOSI score, comparing results preoperatively
Changes in the range of motions | 2, 5 and 10 years follow up.
  Range of motions, comparing postoperative results with preoperative measurements in the operated shoulder

CONTACTS AND LOCATIONS:
Overall Officials: Jon Olav Drogset, MD PhD prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Aalesund Hospital Møre and Romsdal Hospital Trust, Ålesund, Ålesund, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klungsoyr PJ, Guldal F, Vagstad T, Klungsoyr JA. A new subscapular sling operation to stabilize the shoulder. A cadaver study. J Exp Orthop. 2015 Dec;2(1):12. doi: 10.1186/s40634-015-0028-y. Epub 2015 Jun 2. PMID 26914880